CLINICAL TRIAL: NCT03868501
Title: High Working Memory Load to Reduce IGD Cravings: N-Back Task
Brief Title: High Working Memory Load to Reduce Internet Gaming Disorder (IGD) Cravings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, Jin-tao Zhang, Associated Professor, Beijing Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Working memory
Record Dates: First submitted 2019-03-01; First posted 2019-03-11 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Working memory load: n-back task (Experimental): During the intervention, each participant of this group will finish the 3-back task.
  Interventions: Behavioral: n-back task
- Low Working memory load: n-back task (Experimental): During the intervention, each participant of this group will finish the 1-back task.
  Interventions: Behavioral: n-back task

INTERVENTIONS:
Behavioral: n-back task — All participants will be asked to finish the 3-back task and the 1-back task. The 3-back task and the 1-back task will be carried out at intervals to avoid the influence between different tasks. The sequence of the 3-back task and the 1-back task will be counterbalanced across participants.

SUMMARY:
To test whether high working memory load can effectively reduce the craving for IGD.

DETAILED DESCRIPTION:
This project is to use 1-back task and 3-back task to reduce the craving of internet gamers. To test whether high working memory load can effectively reduce the craving for IGD. This project will be conducted in Beijing, China, based on a large sample of internet gamers.

ELIGIBILITY:
Inclusion Criteria:

* The scores of the 9 items of The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition(DSM-5) recommended diagnosis for Internet gaming disorder ≥ 5.
* Engagement in popular Internet games (e.g. Arena of Valor, League of Legends and Player Unknown's Battle Grounds) for over 20 hours per week for a minimum of 12 months.
* The scores of theYoung-Internet Addiction Test(Y-IAT) ≥ 50

Exclusion Criteria:

* Current or history of use of illegal substances and gambling;
* Current or history of psychiatric or neurological illness;
* Current use of psychotropic medications.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-10 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
The craving of internet gamers | 0-1 minutes before each set of cue
  The craving of internet gamers is measured by a single item Visual Analogue Scale with 1 to 7 likert score.
The craving of internet gamers after cue | 0-1 minutes after showing cue
  The craving of internet gamers is measured by a single item Visual Analogue Scale with 1 to 7 likert score.
The craving of internet gamers after tasks | 0-1 minutes after finishing each block of tasks
  The craving of internet gamers is measured by a single item Visual Analogue Scale with 1 to 7 likert score.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tao Zhang, PhD, Study Director — Study Principal Investigator
Locations (1):
- State Key Laboratory of Cognitive Neuroscience and Learning, Beijing Normal University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaag AM, Goudriaan AE, De Vries TJ, Pattij T, Wiers RW. A high working memory load prior to memory retrieval reduces craving in non-treatment seeking problem drinkers. Psychopharmacology (Berl). 2018 Mar;235(3):695-708. doi: 10.1007/s00213-017-4785-4. Epub 2017 Nov 27. PMID 29181814
- [Background] May J, Andrade J, Panabokke N, Kavanagh D. Visuospatial tasks suppress craving for cigarettes. Behav Res Ther. 2010 Jun;48(6):476-85. doi: 10.1016/j.brat.2010.02.001. Epub 2010 Feb 7. PMID 20189549